CLINICAL TRIAL: NCT02241148
Title: Close Kinetic Chain Exercise With Kinesio Taping in the Management of Patellofemoral Pain Syndrome.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Required number of participants were not able to be enrolled.
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, Dr. med. Felix Vilchez Cavazos, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR14-003; OR14-003 (Registry Identifier: closed kinetic chain exercise with kinesio taping); OR14-003 (Registry Identifier: Ejercicios cadena cerrada mas taping); OR14-003 (Other: Universidad Autonoma de Nuevo Leon)
Record Dates: First submitted 2014-07-26; First posted 2014-09-16 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen 500mg (Active Comparator): The control group will receive treatment with acetaminophen 500mg and physical therapy rehabilitation
  Interventions: Drug: Acetaminophen 500mg
- Kinesio taping (Experimental): The experimental treatment group will receive acetaminophen 500mg and physical therapy rehabilitation, plus the application of the technique NUCAP Medical Upper Knee Spider ® Kinesio taping
  Interventions: Device: Kinesio taping

INTERVENTIONS:
Drug: Acetaminophen 500mg — 500 mg, tablets every 8 hours
  Other Names: Tempra® 500mg
  Arms: Acetaminophen 500mg
Device: Kinesio taping — Taping will be changed every week.
  Other Names: SpiderTech ® Kinesio taping
  Arms: Kinesio taping

SUMMARY:
The investigators will include patients attending outpatient clinic in the area of Orthopedics and Traumatology of our hospital with a diagnosis of unilateral Patellofemoral Pain Syndrome.

Two groups would be made, the control group will receive treatment with acetaminophen and physical therapy rehabilitation, closed chain exercises and stretches at home intended for the strengthening of quadriceps, abductors and internal rotators of the hip for the duration of six weeks. The experimental treatment group will receive the above plus the application of the technique NUCAP Medical Upper Knee Spider ® Kinesio taping on the affected knee. Both groups will be evaluated by an external consultation. They will be assessed by the Tegner Activity Scale, the Kujala score of the WOMAC and visual analog scale (VAS) for pain assessment; these scales will be applied at the beginning, third and sixth week

DETAILED DESCRIPTION:
The investigators will include patients attending outpatient clinic in the area of Orthopedics and Traumatology of our hospital with a diagnosis of unilateral Patellofemoral Pain Syndrome. Inclusion criteria are: age between fifteen and thirty-five years, presenting unilateral Patellofemoral pain syndrome with six months of evolution, presenting anterior or retro knee pain that presents itself when undergoing two or more of the following activities: squatting, running, kneeling, jumping, or climbing stairs; physically active patients, with at least thirty minutes of physical activity at least three times per week. Exclusion criteria include patients with previous knee surgeries, chronic pain with more than one year of evolution, pregnancy or suspected pregnancy, application of intra-articular steroids in the three months prior to their evaluation, patients with meniscal injuries, ligament or intra-articular knee structures, degenerative diseases such as diabetes, rheumatoid arthritis, Osteoarthritis of the knee, hip or ankle, history of dislocation or subluxation of patella, Osgood Schlatter syndrome and patellar tendinitis or quadriceps.

The investigators will divide patients into two groups. The control group will receive treatment with acetaminophen and physical therapy rehabilitation, closed chain exercises and stretches at home intended for the strengthening of quadriceps, abductors and internal rotators of the hip for the duration of six weeks. The experimental treatment group will receive the above plus the application of the technique NUCAP Medical Upper Knee Spider ® Kinesio taping on the affected knee. Both groups will be evaluated by an external consultation. They will be assessed by the Tegner Activity Scale, the Kujala score of the WOMAC and visual analog scale (VAS) for pain assessment; these scales will be applied at the beginning, third and sixth week. The patients in the experimental group will be quoted each week to change the tape. The control group will be quoted at the beginning, at three weeks and after six weeks. During the first appointment we will take patients anthropometric measurements (weight, height, BMI) as well as general information. Radiographic studies (anteroposterior and lateral knee, plus the projection Merchant) will be sought to rule out other diseases and see the degree of contact of the patella on the patellofemoral joint. All patients will receive an explanation about their illness, and a booklet with the required exercises as well as their frequency.

For patients to be included in the group of Spider ® Taping, Kinesio Tape pre-cut strips that were placed inferior to the head with no pressure applied, then two bands are placed at the ends of the tape and crossed on the edges of the patella and ending at the thigh to finish applying moderate tension to place them, then two strips were placed at each end of the edges of the first and second tape without applying pressure. The tapes can last up to five days on the extremities while maintaining their purpose, patients included in this group will be summoned each week to remove the tapes and place new ones.

ELIGIBILITY:
Inclusion criteria:

* Age between fifteen and thirty-five years,
* Presenting unilateral PFPS with six months of evolution,
* Presenting anterior or retro knee pain that presents itself when undergoing two or more of the following activities:

(squatting, running,kneeling, jumping,climbing stairs,physically active patients, with at least thirty minutes of physical activity at least three times per week.)

Exclusion criteria:

* Patients with previous knee surgeries,
* Chronic pain with more than one year of evolution,
* Pregnancy or suspected pregnancy
* Application of intra-articular steroids in the three months prior to their evaluation
* Patients with meniscal injuries
* Ligament or intra-articular knee structures
* Degenerative diseases such as diabetes
* Rheumatoid arthritis
* Osteoarthritis of the knee, hip or ankle
* History of dislocation or subluxation of patella
* Osgood Schlatter syndrome
* Patellar tendinitis or quadriceps.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Closed kinetic chain exercise with kinesio taping pain relief measured in the Kujala score | Baseline,3 weeks, 6 weeks
  The Kujala patellofemoral score is a functional evaluation instrument to evaluate knee problems related to the patellofemoral system.It is a 13-item knee-specific self-report questionnaire.
  It documents response to six activities thought to be associated specifically with anterior knee pain syndrome (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp, inability to weight bear through the affected limb, swelling, abnormal patellar movement, muscle atrophy and limitation of knee flexion.

SECONDARY OUTCOMES:
Closed kinetic chain exercise with kinesio taping pain relief measured in the Tegner Activity Scale. | Baseline, 3 weeks, 6 weeks
  The Tegner activity scale was designed as a score of activity level to complement other functional scores for patients with ligamentous injuries. The instrument scores a person's activity level between 0 and 10 where 0 is 'on sick leave/disability' and 10 is 'participation in competitive sports such as soccer at a national or international elite level

OTHER OUTCOMES:
Closed kinetic chain exercise with kinesio taping pain relief measured in WOMAC | Baseline, 3 weeks, 6 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).[2] Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties
Closed kinetic chain exercise with kinesio taping pain relief measured in the visual analog scale (VAS) for pain assessment. | Baseline, 3 weeks, 6 weeks
  The pain VAS is a unidimensional measure of pain intensity. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez, Dr. med., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico